CLINICAL TRIAL: NCT03613441
Title: Impact of Mindful Awareness Practices in Pediatric Residency Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Denise Rita Purdie, MD, FAAP, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001817
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Stress; Burnout, Professional
Keywords: Mindfulness; Residency training
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Awareness Practices (MAPs) (Experimental): Mindful Awareness Practices is a mindfulness-based intervention developed at UCLA's Mindful Awareness Research Center. It is a weekly 2-hour, 6-session, group-based course in mindfulness meditation that is available in-person or online.
  Interventions: Behavioral: Mindful Awareness Practices (MAPs)
- Control (No Intervention): Waitlist control (intervention will be available to this group at the end of the study period)

INTERVENTIONS:
Behavioral: Mindful Awareness Practices (MAPs) — Please refer to arm description
  Arms: Mindful Awareness Practices (MAPs)

SUMMARY:
This study evaluates the effect of a standardized mindfulness based intervention compared to control on self-reported levels of stress in residency trainees.

DETAILED DESCRIPTION:
Recent research studies have indicated that the practice of mindfulness is strongly correlated with enhanced well-being and improved resilience in a variety of populations. Mindfulness-based interventions have been shown to reduce stress and symptoms of burnout in physicians. However, the two studies that included residents were observational trials evaluating the effect of an abbreviated, informal mindfulness course.

The aim of the investigator's study is to assess whether a standardized course in mindfulness meditation (Mindful Awareness Practices, MAPs) reduces self--reported signs and symptoms of stress, burnout, depression, anxiety, loneliness and poor sleep quality in residents in pediatrics training. This study is a randomized controlled trial using 2 parallel groups. The pediatrics residents randomized to the intervention will participate in a standardized mindful awareness practices intervention consisting of one live 45- minute session and 5 web--based self--study sessions. The live session will be administered by a trained mindfulness educator at the UCLA Westwood, Olive View Medical Center and Cedars--Sinai Medical Center campuses. The waitlist group will have the opportunity to participate in the same course once the study has been completed. Participants will respond to questionnaires to assess for levels of stress and other mental health measures before and after the intervention to see if the intervention group had a reduction in symptoms compared to the waitlist group.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric resident at the University of California Los Angeles's Mattel Children's Hospital
* Medicine/Pediatric resident at University of California Los Angeles's Mattel Children's Hospital

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in level of stress per Perceived Stress Scale (PSS) | Baseline and at 2 months (immediately post-intervention)
  PSS = validated 14-item self-report questionnaire of stress experienced over past month. Scores range from 0-56. Higher scores represent a worse outcome.

SECONDARY OUTCOMES:
Change in symptoms of burnout per Abbreviated Maslach Burnout Inventory-9 | Baseline and at 2 months (immediately post-intervention)
  Physician-specific self-report questionnaire of symptoms of burnout. The inventory is divided into three subscales: emotional exhaustion, depersonalization and personal accomplishment. Each subscale scores from 0-18. The subscales are reported separately rather than added together for a total score. Higher scores represent a worse outcome, except on the personal accomplishment subscale, where higher scores represent better outcome.
Change in symptoms of depression per Beck Depression Inventory (BDI) | Baseline and at 2 months (immediately post-intervention)
  Validated self-report questionnaire of symptoms of depression. Scores range from 0-63. Higher scores represent a worse outcome.
Change in symptoms of anxiety per Beck Anxiety Inventory (BAI) | Baseline and at 2 months (immediately post-intervention)
  Validated self-report questionnaire of symptoms of anxiety. Scores range from 0-63. Higher scores represent a worse outcome.
Change in level of loneliness per UCLA Loneliness Scale | Baseline and at 2 months (immediately post-intervention)
  Validated self-report questionnaire of frequency of feeling lonely. Scores range from 20-80. Higher scores represent a worse outcome.
Change in level of sleep quality per Pittsburgh Sleep Quality Index (PSQI) | Baseline and at 2 months (immediately post-intervention)
  Validated self-report questionnaire evaluated sleep quality. Scores range from 0-21. Higher scores represent a worse outcome.
Change in level of mindfulness per Mindful Attention Awareness Scale (MAAS) | Baseline and at 2 months (immediately post-intervention)
  MAAS = validated 15-item self-report questionnaire of tendency to be attentive to and aware of experiences in daily life. Scores range from 15-90. Higher scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Irwin, MD, Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dyrbye L, Shanafelt T. A narrative review on burnout experienced by medical students and residents. Med Educ. 2016 Jan;50(1):132-49. doi: 10.1111/medu.12927. PMID 26695473
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053
- [Background] Irving JA, Dobkin PL, Park J. Cultivating mindfulness in health care professionals: a review of empirical studies of mindfulness-based stress reduction (MBSR). Complement Ther Clin Pract. 2009 May;15(2):61-6. doi: 10.1016/j.ctcp.2009.01.002. Epub 2009 Feb 28. PMID 19341981
- [Background] Romcevich LE, Reed S, Flowers SR, Kemper KJ, Mahan JD. Mind-Body Skills Training for Resident Wellness: A Pilot Study of a Brief Mindfulness Intervention. J Med Educ Curric Dev. 2018 Apr 30;5:2382120518773061. doi: 10.1177/2382120518773061. eCollection 2018 Jan-Dec. PMID 29780891
- [Background] Goldhagen BE, Kingsolver K, Stinnett SS, Rosdahl JA. Stress and burnout in residents: impact of mindfulness-based resilience training. Adv Med Educ Pract. 2015 Aug 25;6:525-32. doi: 10.2147/AMEP.S88580. eCollection 2015. PMID 26347361
- [Derived] Purdie DR, Federman M, Chin A, Winston D, Bursch B, Olmstead R, Bulut Y, Irwin MR. Hybrid Delivery of Mindfulness Meditation and Perceived Stress in Pediatric Resident Physicians: A Randomized Clinical Trial of In-Person and Digital Mindfulness Meditation. J Clin Psychol Med Settings. 2023 Jun;30(2):425-434. doi: 10.1007/s10880-022-09896-3. Epub 2022 Jul 1. PMID 35778655
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860